CLINICAL TRIAL: NCT03508206
Title: Acute Effect of a Standardized Botanical Blend Rich in Polyphenols on Cognitive Functions in Healthy Students: Randomized, Placebo-controlled, Double-blind, Cross-over Clinical Trial
Brief Title: Acute Effect of a Standardized Botanical Blend Rich in Polyphenols on Cognitive Functions in Healthy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Activ'inside (Industry)
Collaborators: CIC SANPSY (USR CNRS 3413), Hôpital Pellegrin, Bordeaux, FRANCE (Unknown); Hospital St André, Bordeaux, FRANCE (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: STUAI2017
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Healthy
Keywords: Students, cognitive functions, memory

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRP arm (Experimental): Food supplement in hard gelatin capsule form containing a Standardized botanical blend rich in polyphenols (SBRP)
  Interventions: Dietary Supplement: SBRP
- Placebo arm (Placebo Comparator): Hard gelatin capsule form containing maltodextrin, with the same appearance as SBRP capsules
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: SBRP — SBRP capsules
  Arms: SBRP arm
Dietary Supplement: PLACEBO — Placebo capsules
  Arms: Placebo arm

SUMMARY:
Available literature suggests that flavanols-rich foods, and more especially monomeric flavanols-rich foods such as grape, can have an acute effect on cognitive functions via different mechanisms such as cerebral blood flow improvement.

The objective of this study is to investigate the effect of a Standardized botanical blend rich in polyphenols (SBRP), on cognitive functions, together with endothelial function in healthy students. Moreover, in order to provide supportive evidence on the mechanisms and biological plausibility to the clinical effects of the product, appropriate biological parameters and circulating metabolites will be assayed.

The study design will be a double-blind, randomised, placebo controlled, crossover study. A total of 30 healthy volunteers will be included. Each participant will receive a single dose of SBRP and placebo capsules, during 2 separate experimental visits and in a counterbalanced order. There will be a 1 week washout period between the 2 experimental visits. During each experimental visit, after a training battery volunteers will be administered a cognitive test battery (COMPASS) before product intake and 6 times after product intake (B1 to B6, from 90 min post-dose to 160 min post-dose).

ELIGIBILITY:
Inclusion Criteria:

* Graduate students (being either at the University or high school), with exam at least every 6 months and attending courses at the equivalent of at least 2 full days each week;
* Male and female subjects (at least 25% of each gender);
* Subjects aged 18 - 25 years (limits included);
* French native speaker;
* Healthy, and especially not suffering from the following diseases, either medically controlled or not:

  * depression,
  * anxiety disorders,
  * diabetes (type I or type II),
  * dyslipidemia,
  * hypertension,
  * any other cardiovascular disease,
  * disorder of the thyroid function.
* Not consuming any food supplements (at time of V0 visit) and agreeing not to consume any food supplements until the end of the study;
* No consumption within the last 30 days (30 days before the V0 visit) of drug or food supplement likely to affect the studied parameters,
* Body Mass Index (BMI) < 30 kg/m2;
* Non-smoker;
* No use of narcotics nor cannabis within the last 7 days (the 7 days preceding the V0 visit) and agreeing not to consume such products until the end of the study. The compliance with this criteria will be confirmed by a urine TetraHydroCannabinol (THC) test at the beginning of the testing visits (V1 and V2);
* Subjects capable of and willing to comply with the protocol and to give their written informed consent.

Exclusion Criteria:

* Exam during the study period;
* Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg during the V0 visit;
* Currently suffering from or personal history of psychiatric or neurologic disorders (examples: schizophrenia, depression, generalized anxiety disorder, epilepsia) according to the subject's self-declaration;
* Neuroleptic, hypnotic, anxiolytic or antidepressant treatment (whatever the reason) ongoing or stopped since less than 3 months;
* Anti-hypertensive, blood thinner or anticoagulant treatment (eg aspirin > 325mg / day and prescribed as anticoagulant) ongoing or stopped since less than 3 months;
* Venotonic treatment or vasodilator treatment ongoing or stopped since less than 3 months;
* Any other treatment (administered systemically or locally) that may affect the endothelial function (example: statins);
* History of moderate to severe traumatic brain injury and / or intracranial surgery;
* Personal history of Cerebrovascular Accident (CVA);
* Inflammatory bowel disease (examples: Crohn disease, coeliac disease, irritable bowel syndrome) likely to affect the intestinal absorption of the study product components;
* Progressive disease ongoing or resolved since less than one year;
* General anesthesia in the last 7 days or planned in the next 2 weeks;
* Restrictive or unbalanced diet (hypocaloric diet aiming at weight loss, vegan, …) according to the subject's self-declaration at V0;
* Excessive alcohol consumption : more than 2 glasses per day every day;
* Documented food allergy to one of the components of the study product;
* Psychological or linguistic incapability to sign the informed consent;
* Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* Participation in another biomedical study or during the exclusion period of a previous study;
* Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in the number of correct answers during the Serial Three Subtraction task (Serial Three) between the baseline battery and the 4th repetition of the battery after product intake (B4). | From baseline to 120 min post-dose
  The Serial Three task will be administered through the computerized COMPASS battery (" Computerised Mental Performance Assessment System "). Serial subtraction tasks rely on working memory (executive function).

SECONDARY OUTCOMES:
Changes in the number of correct responses from the Serial Three Subtraction task between the baseline battery and each of the repetitions N°1, 2, 3, 5 and 6 of the battery after product intake | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the number of correct responses from the Serial Three Subtraction task between the first repetition after product intake and the repetitions N°2 to 6 | From 90 to 160 min post-dose
  Differences between the values obtained during the first post-dose battery and the next repetitions;
Changes in the number of errors from the Serial Three Subtraction task (Serial Three, COMPASS battery) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the number of correct responses from the Serial Sevens Subtraction task (Serial Sevens, COMPASS battery) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the number of errors from the Serial Sevens Subtraction task (Serial Sevens, COMPASS battery) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the reaction time from the RVIP test (" Rapid Visual Information Processing ", COMPASS battery), in milliseconds (ms) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the percentage of correct responses from the RVIP test (COMPASS battery) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the number of false alarms from the RVIP test (COMPASS battery) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the score of mental fatigue (COMPASS battery self-assessment using a Visual Analogue Scale) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the score of anxiety (COMPASS battery, VAS) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the score of vigilance/ alertness (COMPASS battery, VAS) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Changes in the score of cognitive performances (COMPASS battery, VAS) between the baseline battery and each of the repetitions of the battery after product intake (B1 to B6); | From baseline to 160 min post-dose
  Differences between each battery and baseline values;
Number of correct responses at the immediate free recall test before the first repetition of the test battery (B1) ; | 85-90 min post-dose
  Number of words properly recalled, among a list of 20 words, with no clue
Number of correct responses at the delayed free recall test, after the last repetition of the test battery (B6) ; | 165-170 min post-dose
  Number of words properly recalled, among a list of 20 words, with no clue
Number of correct responses at the delayed recognition task, after the last repetition of the test battery (B6) ; | 165-170 min post-dose
  Number of words properly recognized among a list of 20 words containing 10 words from the original list and 10 distractors
Changes between the values measured in fasting conditions and those measured after the end of the cognitive assessments in flow-mediated dilation (FMD) | Before product administration; 180 min post-dose
  Post-ischemic increase of brachial artery diameter, in % of the pre-ischemic diameter
Changes between the values measured in fasting conditions and those measured after the end of the cognitive assessments (i.e. 3 hours after product intake) in basal diameter of brachial artery; | Before product administration; 180 min post-dose
  Pre-ischemic diameter of brachial artery (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- SANPSY (CHU Pellegrin), Bordeaux, France

IPD SHARING:
Plan to Share IPD: No